CLINICAL TRIAL: NCT07331844
Title: The Combined Effect of Botulinum Toxin Type A and Mirror Therapy in the Management of Chronic-Phase Upper Extremity Spasticity After Ischemic Stroke: A Double-Blind, Controlled Study
Brief Title: BTX-A and Mirror Therapy for Chronic Stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSM AYNA BOTULİNUM
Record Dates: First submitted 2025-02-25; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Spastic Hemiplegia
Keywords: STROKE; MİRROR THERAPY; BOTULİNUM TOXİNS
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Botulinum Toxins, Type A; Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BTX-A and MİRROR THERAPY (Active Comparator): Participants were asked to sit in a chair and place both forearms on an exercise table with their elbows flexed at 90 degrees. To administer mirror therapy, the direct view of both the healthy and the hemiplegic hand and wrist was blocked using a partition method. A mirror was then placed between the two forearms, ensuring that the mirror image of the healthy-side wrist overlapped with the position of the hemiplegic-side wrist. By observing the healthy hand's movements through the mirror during the exercises, a visual movement illusion was created for the hemiplegic hand.
  Interventions: Drug: Botulinum toxin type A (Botox®, Allergan); Procedure: Mirror Therapy
- BTX-A + Sham Mirror Therapy (Active Comparator): In the sham group, however, a transparent glass was used instead of a mirror, and participants were asked to watch the wrist movements of the paralyzed side through the glass, providing visual feedback without creating an illusion. The sham procedure was applied for the same duration using the transparent glass
  Interventions: Drug: Botulinum toxin type A (Botox®, Allergan); Procedure: Sham Mirror Therapy

INTERVENTIONS:
Drug: Botulinum toxin type A (Botox®, Allergan) — Botulinum toxin type A was administered via intramuscular injections into the spastic upper limb muscles based on clinical evaluation. Injection sites and dosages were individualized according to the distribution and severity of spasticity. All injections were performed prior to the rehabilitation interventions.
Procedure: Mirror Therapy — Mirror therapy was performed with participants seated and both forearms placed on a table. A mirror was positioned between the limbs to create a visual illusion of movement of the affected limb by observing the movements of the unaffected limb.
  Arms: BTX-A and MİRROR THERAPY
Procedure: Sham Mirror Therapy — Sham mirror therapy was performed using a transparent glass panel instead of a mirror, allowing visual feedback without inducing a mirror illusion. Session frequency and duration were identical to those of the mirror therapy group.
  Arms: BTX-A + Sham Mirror Therapy

SUMMARY:
Stroke is one of the leading causes of disability worldwide, particularly affecting the upper extremities and thus negatively impacting patients' activities of daily living and quality of life. Upper extremity spasticity, characterized by increased muscle tone and tendon reflexes, leads to functional limitations. While Botulinum Toxin Type A (BTX-A) is widely used to manage spasticity and can temporarily alleviate symptoms, it does not directly support neuroplasticity and often requires repeated injections.

Mirror therapy (MT) has emerged as a promising rehabilitation approach with the potential to stimulate motor recovery and cortical reorganization. It is hypothesized that combining MT with BTX-A injections may more effectively reduce spasticity and improve upper extremity function.

In this study, a randomized, sham-controlled, double-blind, prospective design was employed to investigate the effects of adding MT to BTX-A treatment on spasticity and upper extremity motor function in stroke patients. A total of 30 patients, who received BTX-A injections, were divided into two groups: an experimental group receiving mirror therapy and a control group receiving sham therapy (using transparent glass). All patients also underwent a standardized conventional rehabilitation program, and the BTX-A injection protocol was kept consistent. Treatment efficacy was evaluated by comparing pre-injection measurements with those at six months post-injection, using the Brunnstrom Scale, Modified Ashworth Scale (MAS), Fugl-Meyer Scale, and a hand dynamometer. The findings are expected to shed light on the potential benefits of simultaneous MT and BTX-A administration, including reducing injection frequency, and to guide more comprehensive approaches in the rehabilitation of chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of unilateral ischemic stroke
* Under the routine medical follow-up of the same clinician who plans upper extremity BTX treatment based on standard medical indications
* At least 3 months post-stroke
* Signed informed consent form
* Mini-Mental State Examination (MMSE) score >24
* Fugl-Meyer Assessment score <55
* Modified Ashworth Scale (MAS) score of 1-4

Exclusion Criteria:

* Any prior BTX-A or other injections administered to the upper extremity Severe cognitive impairment or any mental disorder preventing effective communication
* Concurrent enrollment in another experimental treatment program
* Visual or motor deficits that would prevent the application of mirror therapy
* History of multiple strokes
* Presence of neuromuscular pathology in the unaffected extremity
* Stroke due to a non-ischemic cause

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
FUGL MAYER SCORE | 6 MONTH
  The Fugl-Meyer Motor Section focuses on evaluating the motor functions of the upper and lower extremities in individuals who have had a stroke. The tests in this section are scored based on fundamental parameters such as muscle activity, synergy patterns, joint movement control, and coordination. The total motor score commonly reaches 66 points (although there are versions with different point ranges). A higher Fugl-Meyer Motor Section score reflects better motor function in the individual.

SECONDARY OUTCOMES:
ASHWORTH SCALE | 6 MONTH
  The Ashworth Scale is a clinical measurement tool used to objectively evaluate the level of spasticity. The scale is scored from 0 to 4 (including 1+). The higher the score, the greater the resistance to passive movement (indicating more pronounced spasticity)
BRUNNSTROM LEVEL | 6 MONTH
  Brunnstrom evaluates the upper extremity and the hand separately in six fundamental stages. The upper extremity staging assesses synergy and movement capabilities of the shoulder, elbow, and wrist. The hand staging reflects the ability to grasp, release, and perform fine motor skills. As the stages advance over time (for example, progressing from Stage 3 to Stage 4), the effectiveness of rehabilitation and the patient's recovery process are monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Liv hospital Vadistanbul, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT07331844/Prot_SAP_000.pdf